CLINICAL TRIAL: NCT01404442
Title: Evaluation of the Analgesic Effect of Midazolam and Ketamine as an Additive to Intrathecal Bupivacaine in Patients Undergoing Cesarean Section
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, marzieh beigom khezri, Assistant professor, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACTRN12611000729921
Record Dates: First submitted 2011-07-21; First posted 2011-07-28 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Post Operative Pain
Keywords: midazolam; ketamine; intrathecal; pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ketamine (Active Comparator): The ketamine group (groupK) received bupivacaine 10mg combined with 0.1 mg/kg ketamine preservative free intrathecally .
  Interventions: Drug: Ketamine
- midazolam (Active Comparator): The midazolam group (group M) received bupivacaine 10mg combined with0.02 mg/ kg midazolam intrathecally
  Interventions: Drug: Midazolam
- placebo (Placebo Comparator): The placebo group (group P) received bupivacaine 10mg combined with 0.5ml distilled water intrathecally .
  Interventions: Drug: placebo(distilled water

INTERVENTIONS:
Drug: placebo(distilled water — The placebo group (group P) received bupivacaine 10mg combined with 0.5ml distilled water intrathecally .
  Arms: placebo
Drug: Ketamine — The ketamine group (groupK) received bupivacaine 10mg combined with 0.1 mg/kg ketamine preservative free intrathecally
  Arms: Ketamine
Drug: Midazolam — The midazolam group (group M) received bupivacaine 10mg combined with0.02 mg/ kg midazolam intrathecally
  Arms: midazolam

SUMMARY:
Objective :To compare the analgesic effect of intrathecal midazolam and ketamine as an additive to bupivacaine in patients undergoing cesarean section .

Methods:Following Ethics Committee approval and informed patients consent, Ninety patients 18-45 yr old ASA physical status I or II, scheduled for cesarean section under spinal anesthesia, were studied in a prospective, double-blinded, randomized way. The patients were randomly allocated to one of three groups of 30 each. The ketamine group (groupK) received bupivacaine 10mg combined with 0.1 mg/kg ketamine preservative free ,the midazolam group (group M) received bupivacaine 10mg combined with0.02 mg/ kg midazolam and the placebo group (group P) received bupivacaine 10mg combined with 0.5ml distilled water intrathecally . Time to first requirement of analgesic supplement, Sensory block onset time, maximum sensory level , onset of motor block, duration of blockade, hemodynamics variables, the incidence of hypotension, ephedrine requirements, bradycardia ,hypoxemia [Saturation of peripheral oxygen (SpO2)<90], postoperative analgesic requirements and Adverse events, such as sedation, dizziness , Pruritus and postoperative nausea and vomiting were recorded. Patients were instructed preoperatively in the use of the verbal rating scale (VRS) from 0 to 10 (0no pain, 10maximum imaginable pain) for pain assessment. If the VRS exceeded four and the patient requested a supplement analgesic, diclofenac Na supp 100 mg was to be given for post-operative pain relief as needed . For breakthrough pain(VRS >4) if time of administration of diclofenac Na less than 8h,Pethidine 25 mg IV was given.

DETAILED DESCRIPTION:
The patients were randomly allocated to one of three groups of 30 each. The ketamine group (groupK) received bupivacaine 10mg combined with 0.1 mg/kg ketamine preservative free ,the midazolam group (group M) received bupivacaine 10mg combined with0.02 mg/ kg midazolam and the placebo group (group P) received bupivacaine 10mg combined with 0.5ml distilled water intrathecally .

ELIGIBILITY:
Inclusion Criteria:

* patients with American Society of Anesthesiologists(ASA) physical status I and II, undergoing elective cesarean section

Exclusion Criteria:

* significant coexisting disease such as hepato-renal and cardiovascular disease
* any contraindication to regional anesthesia such as local infection or bleeding disorders
* allergy to ketamine or midazolam
* long-term opioid use or a history of chronic pain.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Time to first requirement of analgesic supplement | participants will be followed for the duration of 24 hours after intratechal injection (Time from the injection of intrathecal anesthetic solution to first requirement of analgesic supplement will be recorded.)
  analgesic administration was initiated by patient request(verbal rating scale[ VRS]>4)
Postoperative analgesic requirements | 24 hours postoperative(Time from the injection of intrathecal anesthetic solution to 24 hours postoperative)
  postoperative analgesic requirements will be assessed by verbal rating scale (VRS) from 0 to 10 (0no pain, 10maximum imaginable pain).Each administration was initiated by patient request( VRS>4)

SECONDARY OUTCOMES:
Sensory block onset time will be assessed by a pinprick test | sensory block will be assessed by pinprick test every 10 seconds following intrathecal injection
  The onset of sensory block was defined as the time between the end of injection of the intrathecal anesthetic and the absence of pain at the T10 dermatome
duration of sensory block will be assessed by a pinprick test | sensory block will be assessed by pinprick test every 5 minuts following intrathecal injection
  The duration of sensory block was defined as the time for regression from the maximum block height sensory block to T10 dermatom will be assessed by pinprick test every 5 minuts following intrathecal injection
the onset of motor block will be assessed by the modified Bromage score | every10 seconds following intrathecal injection
  The onset of motor block was defined as the time between the end of injection of the intrathecal anesthetic to Bromage block 1
hemodynamic variables are assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 5min before the intrathecal injection
hemodynamic variables are assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 2minutes after intrathecal injection
hemodynamic variables are assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 4minutes after intrathecal injection
hemodynamic variables are assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 6minutes after intrathecal injection
hemodynamic variables are assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 8minutes after intrathecal injection
hemodynamic variables are assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 10 minutes after intrathecal injection
hemodynamic variables are assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 15minutes after intrathecal injection
hemodynamic variables are assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 20 minutes after intrathecal injection
hemodynamic variables are assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 25 minutes after intrathecal injection
hemodynamic variables are assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 30 minutes after intrathecal injection
duration of motor block will be assessed by the modified Bromage score | every 5 minutes following intrathecal injection
  duration of motor block was defined the time from intrathecal injection to Bromage score0

CONTACTS AND LOCATIONS:
Overall Officials: Marzieh Beigom Khezri, Principal Investigator — Qazvin medical science university
Locations (1):
- Qazvin university of medical science, Qazvin, Qazvin Province, Iran

REFERENCES:
- [Derived] Khezri MB, Ghasemi J, Mohammadi N. Evaluation of the analgesic effect of ketamine as an additive to intrathecal bupivacaine in patients undergoing cesarean section. Acta Anaesthesiol Taiwan. 2013 Dec;51(4):155-60. doi: 10.1016/j.aat.2013.12.004. Epub 2014 Jan 21. PMID 24529671